CLINICAL TRIAL: NCT01926366
Title: A Randomized, Double-Blind, Third-Party-Unblinded, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of AZD6423 in Healthy Volunteers
Brief Title: AZD6423 SAD/MAD Study in Healthy Volunteers
Acronym: AZD6423
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3521C00001
Record Dates: First submitted 2013-08-12; First posted 2013-08-20 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: AZD6423 (Experimental): Subjects will participate in 1 of 8 groups and receive single or multiple doses of AZD6423 or matching placebo. In each group 6 subjects will receive AZD6423 and 2 subjects will receive matching placebo.
  Interventions: Drug: AZD6423
- Placebo to match AZD6423 (Placebo Comparator): Subjects will participate in 1 of 8 groups and receive single or multiple doses of AZD6423 or matching placebo. In each group 6 subjects will receive AZD6423 and 2 subjects will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6423 — Drug: AZD6423 Single or Multiple doses via infusion.
  Arms: Experimental: AZD6423
Drug: Placebo — Placebo to match AZD6423 Single or Multiple doses of matching placebo delivered via infusion
  Arms: Placebo to match AZD6423

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of single and multiple ascending dosage levels of AZD6423 in healthy volunteers. The study includes an up to 28-day screening period, an in-house period during which AZD6423 or placebo will be administered IV, and a 4- to 10-day follow-up period after discharge.

DETAILED DESCRIPTION:
In Part 1 of the study (single ascending dose portion), approximately 40 subjects will be randomly assigned. Eight (8) subjects will be randomized in each of 5 dosage-level cohorts (AZD6423 or placebo). Within each cohort, 6 subjects will be randomized to receive AZD6423 and 2 subjects will be randomized to receive placebo. Each subject will receive only one dose of either AZD6423 or placebo on Day 1. In Part 2 of the study (multiple ascending dose portion), approximately 24 subjects will be randomly assigned. Eight (8) subjects will be randomized in each of 3 dosage-level cohorts. Within each cohort, 6 subjects will be randomized to receive AZD6423 and 2 subjects will be randomized to receive placebo. Each subject will receive three doses of either AZD6423 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand the nature of the study and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-specific procedures.
2. All male subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control for the duration of the study and for 15 days after dose administration. A male subject is considered biologically capable of having children even if his sexual partner is sterile or using contraceptives.
3. Subjects must have a body mass index (BMI) between 19 and 30, inclusive and weigh between 50kg and 100kg inclusive.
4. Subjects must be fluent in English.

Exclusion Criteria:

1. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality.
2. A clinically significant abnormality on physical examination, neurological examination, EEG, ECG, vital signs or laboratory evaluations at screen or between screen and dose administration.
3. A history of seizure.
4. A history of head trauma, including closed head injury with loss of consciousness.
5. Any history of suicide attempt or suicidal behavior, or, in the opinion of the investigator, clinically significant risk of suicide or violent behavior.
6. Urine drug screen positive for a drug of abuse
7. A family history of schizophrenia, schizoaffective disorder, or psychosis in first degree relatives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of AZD6423 in healthy subjects via adverse events | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via EEG | From Baseline up to 6 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via ECG. | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via vital signs (blood pressure and pulse). as well as body temperature and weight | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via clinical laboratory tests (chemistry, hematology and urinalysis). | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via psychiatric assessments. | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via neurological exams. | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.
Assessment of the safety and tolerability of AZD6423 in healthy subjects via physical exams. | From Baseline up to 18 days
  The primary objectives of this study are to assess the safety and tolerability of single and multiple ascending dosage levels of AZD6423 versus placebo in healthy volunteers.

SECONDARY OUTCOMES:
Description of the PK profile for AZD6423 in terms of: observed maximum plasma concentration (Cmax), time to reach maximum plasma concentration (tmax), terminal rate constant (λz), terminal half-life (t½ z), and area under the curve (AUC). | From Baseline up to 7 days
  Secondary objectives are to assess the pharmacokinetics and pharmacodynamics of AZD6423 in healthy volunteers.
Assessment of the pharmacodynamics of AZD6423 in terms of the relationship between plasma concentration of AZD6423 and EEG | From Baseline up to 7 days
  Secondary objectives are to assess the pharmacokinetics and pharmacodynamics of AZD6423 in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D., Principal Investigator — California Clinical Trials
Locations (1):
- Research Site, Glendale, California, United States